CLINICAL TRIAL: NCT03505827
Title: Visual Field Changes in Patients Undergoing TECNIS ZCB00 Monofocal vs. TECNIS Symfony Extended Depth of Focus Intraocular Lens Implantation
Brief Title: Visual Field Changes in TECNIS ZCB00 Monofocal vs. TECNIS Symfony Extended Depth of Focus Intraocular Lens Implantation
Status: Withdrawn | Type: Observational
Why Stopped: No participants were successfully enrolled.
Sponsor: Western University, Canada (Other)
Collaborators: Ivey Eye Institute (Other)
Responsible Party: Principal Investigator, Tony Lin, Principal Investigator, Western University, Canada
Other Study IDs: 111201
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Lenses, Intraocular; Visual Fields; Cataract
Keywords: TECNIS Symfony
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TECNIS Monofocal: This group of patients has chosen to undergo implantation of a TECNIS monofocal ZCB00 lens during cataract surgery. This decision was made prior to enrolment in the study. This group of patients will receive standard of care cataract surgery, as any other patient would. The sole intervention we will be undertaking is a 24-2 Humphrey visual field test prior to surgery, and a 24-2 SITA standard Humphrey visual field test after surgery at 1 month post-operatively.
  Interventions: Diagnostic Test: 24-2 SITA Standard Humphrey Visual Field Test
- TECNIS Symfony: This group of patients has chosen to undergo implantation of a TECNIS Symfony extended depth of focus lens during cataract surgery. This decision was made prior to enrolment in the study. This group of patients will receive standard of care cataract surgery, as any other patient would. The sole intervention we will be undertaking is a 24-2 SITA standard Humphrey visual field test prior to surgery, and a 24-2 Humphrey visual field test after surgery at 1 month post-operatively.
  Interventions: Diagnostic Test: 24-2 SITA Standard Humphrey Visual Field Test

INTERVENTIONS:
Diagnostic Test: 24-2 SITA Standard Humphrey Visual Field Test — Patients participate in a 24-2 SITA Standard humphrey visual field test. This includes sitting in a dark room at a visual field machine. Stimulus test points of different intensity and size will be presented to the patient, as per SITA standard protocol. The patient will indicate by pressing a button when they see the visual stimulus.

SUMMARY:
Glaucoma is a leading cause of blindness worldwide. Damage to the optic nerve results in vision loss gradually. This vision loss can be detected by using visual field testing, and is a way of monitoring glaucoma progression. As this population ages, cataracts develop, and patients need to undergo cataract surgery to replace the cloudy crystalline lens with an artificial intraocular lens (IOL). The standard of treatment is implantation of a monofocal IOL, but this limits depth of focus and does not allow clear vision at both distance and near without glasses post-operatively. Multifocal and trifocal lenses split light into multiple distinct foci at near, intermediate and far distances without glasses correction. However, these lenses have been shown to reduce contrast sensitivity and impair visual field testing results, and are not recommended in patients with glaucoma. The TECNIS Symfony IOL has recently been approved by Health Canada and offers an extended range of vision with a single elongated focal point to allow patients to see at both distance and near. The lens is advertised to enhance contrast sensitivity, but it is currently unknown whether the TECNIS Symfony IOL impacts visual field testing. We will study the visual field changes in patients undergoing both TECNIS ZCB00 monofocal and TECNIS Symfony extended depth of focus IOL implantation during cataract surgery. The results of this study will impact the advice cataract surgeons give to patients with glaucoma, regarding whether this population of patients would benefit from a standard monofocal IOL implantation or an extended depth of focus TECNIS Symfony IOL implantation.

DETAILED DESCRIPTION:
Primary open angle glaucoma is a leading cause of blindness worldwide, and is the most common form of glaucoma. This condition involves progressive damage to the optic nerve over time and ultimately vision loss that can be detected using standard automated perimetry visual field testing. As this population ages, patients will eventually develop cataracts and require cataract surgery to replace the cloudy crystalline lens with an artificial intraocular lens. The standard of treatment is implantation of a monofocal intraocular lens (IOL), but this limits depth of focus and does not allow clear vision at both distance and near without spectacle correction post-operatively. To provide a refractive component to cataract surgery, multifocal and trifocal lenses were introduced and split light into multiple distinct foci at near, intermediate and far distances without correction. However, splitting of incoming light has the potential to decrease contrast sensitivity and increase photic phenomena. In addition, multifocal IOLs have been shown to reduce mean deviation on automated perimetry compared to monofocal IOLs and are not recommended in patients where visual field reduction may not be tolerated, such as in patients with glaucoma. The TECNIS Symfony IOL has been recently been approved by Health Canada and offers extended range of vision with a single elongated focal point, corrects for chromatic aberration and results in contrast enhancement. It is unknown whether this new IOL impacts visual field testing in glaucoma patients post cataract surgery.

The objective of this study is to compare visual field outcomes in patients choosing to undergo cataract surgery with either a TECNIS ZCB00 monofocal vs TECNIS Symfony extended depth of focus intraocular lens.

It is hypothesized that patients who undergo implantation of a TECNIS Symfony extended depth of focus intraocular lens will have impaired visual field testing (a decrease in mean deviation on Humphrey 24-2 standard automated perimetry) compared to those undergoing TECNIS ZCB00 monofocal intraocular lens implantation.

This will be a prospective cohort study.

Patients undergoing either TECNIS ZCB00 monofocal or TECNIS Symfony extended depth of focus ZXR intraocular lens insertion during cataract surgery will be recruited.

Patients will not be approached regarding the study until the patient decides which lens will be inserted during surgery. This study has no impact on a patient's choice of intraocular lens. This study will not be assigning a lens as part of the intervention.

There will be no randomization of the groups, given that patients will be choosing which lens will be implanted during surgery pre-operatively, as any other patient undergoing cataract surgery would.

There will be no blinding of study participants or of the investigators.

As per standard pre-operative assessment, patients will have ocular Biometry performed prior to surgery to assess what prism diopter lens to insert intra-operatively.

On the day of this appointment, participants will be asked to perform a 24-2 Humphrey standard automated perimetry visual field test with Swedish Interactive Threshold Algorithm (SITA) standard thresholds.

In addition, at the 1-month post-operative appointment, participants will be asked to again complete a 24-2 Humphrey visual field, in addition to the standard post-operative examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chosen to undergo elective cataract surgery in one eye with 20/40 - 20/100 vision (best corrected) in the operated eye on initial pre-op surgical assessment and with greater than or equal to 20/25 vision (best corrected) in the operated eye at 1-month post-operatively.
* Patients who have chosen to undergo TECNIS ZCB00 monofocal intraocular lens implantation.
* Patients who have chosen to undergo implantation of a TECNIS Symfony extended depth of focus intraocular lens.
* Patient must be able to reliably perform visual field testing.
* No other eye disease other than cataract.
* Patient must be older than 18 years of age.
* Patient must be proficient in the English language.

Exclusion Criteria:

* Patients who are unwilling or unable to undergo visual field testing.
* Patients with glaucoma.
* Patients who have history of laser refractive surgery.
* Patients who experienced an intra-operative complication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patients undergoing cataract surgery at the Ivey Eye Clinic in London, Ontario, Canda who chose to receive a TECNIS Symfony intraocular lens implant or TECNIS monofocal ZCB00 intraocular lens implant will be approached to be enrolled in the study AFTER determining their decision to undergo cataract surgery and decision of lens implantation has been made.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Mean Deviation | 1 year
  An overall value of the total amount of visual field loss

SECONDARY OUTCOMES:
Pattern Standard Deviation | 1 year
  The sum of the absolute value of the difference between the threshold value for each point and the average visual field sensitivity at each point.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lin, MD, Principal Investigator — Western University
Locations (2):
- Canada (2):
  - Ivey Eye Institute, London, Ontario
  - St. Joseph's Health Care London, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farid M, Chak G, Garg S, Steinert RF. Reduction in mean deviation values in automated perimetry in eyes with multifocal compared to monofocal intraocular lens implants. Am J Ophthalmol. 2014 Aug;158(2):227-231.e1. doi: 10.1016/j.ajo.2014.04.017. Epub 2014 Apr 29. PMID 24784872
- [Background] de Medeiros AL, de Araujo Rolim AG, Motta AFP, Ventura BV, Vilar C, Chaves MAPD, Carricondo PC, Hida WT. Comparison of visual outcomes after bilateral implantation of a diffractive trifocal intraocular lens and blended implantation of an extended depth of focus intraocular lens with a diffractive bifocal intraocular lens. Clin Ophthalmol. 2017 Oct 26;11:1911-1916. doi: 10.2147/OPTH.S145945. eCollection 2017. PMID 29138533
- [Background] Shen Z, Lin Y, Zhu Y, Liu X, Yan J, Yao K. Clinical comparison of patient outcomes following implantation of trifocal or bifocal intraocular lenses: a systematic review and meta-analysis. Sci Rep. 2017 Mar 28;7:45337. doi: 10.1038/srep45337. PMID 28422087
- [Background] Nouri-Mahdavi K. Selecting visual field tests and assessing visual field deterioration in glaucoma. Can J Ophthalmol. 2014 Dec;49(6):497-505. doi: 10.1016/j.jcjo.2014.10.002. PMID 25433738
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815